CLINICAL TRIAL: NCT02957006
Title: Discrimination of P and T-waves With Linq and Holter
Brief Title: Discrimination of P and T Waves With Linq and Holter
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TriHealth Inc. (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-120
Record Dates: First submitted 2016-11-04; First posted 2016-11-07 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Loop Recorder — Observation of Loop Recorder implanted for clinical reasons

SUMMARY:
Currently loop recorders diagnose arrhythmias and send automatic alerts to physicians based on R to R relationships only. We believe arrhythmia diagnostics could be improved if accurate detection of P and T waves as well as QRS complexes were possible.

There is no technique available for long term outpatient monitoring of QT intervals for patient at risk of torsade de pointes when receiving QT prolonging drugs. We believe that if an accurate T wave detection algorithm were developed loop recorders could be used to monitor the QT interval, and perhaps even provide alerts for patients at risk.

The objective of this study is to see if an algorithm can be developed to accurately define P and T waves using data from an implantable loop recorder.

DETAILED DESCRIPTION:
Pilot Study of 20 prospective cardiology patients with loop recorders currently implanted for standard clinical indications.

Eligible Subjects will be brought into the office of John Wilson, MD or Marshall Winner, MD. After informed consent is obtained from Hatton Research Staff the following will be performed:

* subjects will have an initial loop recorder download to USB flash drive
* 12 lead EKG
* Annotated QT intervals on a 30 second rhythm strip
* 24 hour Holter monitor placed by Hatton Research Staff in order to confirm the loop recorder data.
* Subjects will be instructed on the Holter monitors care and use.
* Subjects will be scheduled to come back to the office after 24 hours to return the Holter monitor and have a final loop recorder download completed.
* Data from the loop recorder, Holter monitor, 12 lead EKG, and 30 second rhythm strip will be downloaded and de-identified per Hatton Research Staff.
* All de-identified data from the initial loop recorder download, 12 lead EKG, 30 second rhythm strip, final loop recorder download, and Holter monitor will be sent to Medtronic for algorithm development.

Independent Variables: These variables include age and race Dependent Variables: These variables include the data from the loop recorder, 12 lead EKG, Holter monitor and 30 second rhythm strip.

Intervention or experimental aspect of the study Subjects will have a 12 lead EKG performed with 30 second rhythm strip Subjects will complete a period of 24 hours in which they will wear a Holter monitor applied by Hatton Research Staff.

Statistical Analysis

* Descriptive statistics (mean, standard deviation) will be calculated for all continuous variables. Continuous variables will be compared using Student's - T test or ANOVA as appropriate.
* Frequency and percentages will be calculated for all categorical variables.
* Categorical data will be compared using chi square or Fisher's Exact Test as appropriate
* Data variables will be assessed by Hatton Research Specialist

ELIGIBILITY:
Inclusion Criteria:

* Subject currently has a Medtronic loop recorder implanted
* Subject has large enough P and T wave amplitudes present per discretion of MD.

Exclusion Criteria:

* Subjects with inadequate sized P and T waves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who currently have a loop recorder implanted
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
If an accurate algorithm to detect P and T waves along with QRS recognition were developed implantable loop recorders arrhythmia diagnostic capabilities could be improved and expanded. This study will collect data for the development of such algorithms. | Data analysis will be completed 1-2 months after enrollment complete

CONTACTS AND LOCATIONS:
Overall Officials: John Wilson, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No